CLINICAL TRIAL: NCT03015766
Title: Auricular Acupressure for Hemodialysis Patients With Insomnia: Study Protocol for a Multi-centre Double-blind, Randomized Controlled Trial
Brief Title: Auricular Acupressure for Hemodialysis Patients With Insomnia
Acronym: AAHDIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Qizhan Lin, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YN2015MS25
Record Dates: First submitted 2016-12-22; First posted 2017-01-10 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Insomnia Chronic
Keywords: insomnia; hemodialysis; auricular acupressure; randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupressure therapy (Experimental): Participants in the treatment group will received AAT on five active acupoints including Acup.1. Shen Men (Spiritual Gate, TF4), Acup.2. Jiao Gan (Sympathetic autonomic, AH6a), Acup.3. Xin (Heart, CO15), Acup.4. Pi Zhi Xia (Subcortex, AT4), Acup.5. Nei Fen Mi (Endocrine, CO18)
  Interventions: Other: auricular acupressure therapy
- sham auricular acupressure therapy (Sham Comparator): Participants in the control group (SAA group) will receive auricular acupressure on five Helix points (HX 5-9), which were clearly remote from the inner ear area. These points have no evidence for insomnia management.
  Interventions: Other: sham auricular acupressure therapy

INTERVENTIONS:
Other: auricular acupressure therapy — Auricular acupressure, is a therapeutic method in which specific acupoints on the ear are stimulated to treat various disorders of the body. This practice is based on the theory that there are specific points on the auricle which correspond to major organs or systems of the body; and therapeutic effect on the corresponding target organ or system can be exerted by manipulating auricular acupoints. Auricular acupressure applies stimulation through pressure on specific acupoints by the imbedded beads, usually Semen Vaccaria (Wang Bu Liu Xing) or stainless steel beads. This therapeutic method is non-invasive and can be self-manipulated by the recipients at times required.
  Other Names: auricular acupressure; ear acupressure
  Arms: Auricular acupressure therapy
Other: sham auricular acupressure therapy — The intervention is the same as that in the experimental group only when the points are five Helix points (HX 5-9). These points are clearly remote from the inner ear area and have no evidence for insomnia treatment.
  Other Names: sham AAT
  Arms: sham auricular acupressure therapy

SUMMARY:
Auricular acupressure therapy (AAT) has been applied in MHD patients with insomnia in recent years and yielded favorable results. However, the effect and safety of AAT for insomnia in MHD population still lacks high quality evidence. A randomized controlled clinical trial is planned to evaluate the effect and safety of AAT in MHD patients with insomnia.

DETAILED DESCRIPTION:
Insomnia, a worldwide health problem, is much more frequently complained in maintenance hemodialysis (MHD) patients and impairs their quality of life and long term outcome. Hypnotic sedative agents are often reluctantly prescribed with doses mounting up. Patients are concerned about drug dependence and drug-related adverse effects. As a non-drug therapy, auricular acupressure therapy (AAT) is attractive to both patients and practitioners and is widely used to treat many conditions in China. The investigators had been applying AAT for MHD patients with insomnia in recent years and yielded favorable results. However, the effect and safety of AAT for insomnia in MHD population still lacks high quality evidence. Therefore, the investigators aimed to perform a randomized controlled clinical trial in MHD patients with insomnia to evaluate the effect and safety of AAT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18~75 years
* On regular dialysis ( 2 - 3 sessions weekly, 4 hours each session, total weekly dialysis hours ≥ 10 hours) for more than 3 months (but less than 10 years)
* Insomnia according to The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Global score of PSQI > 7
* Informed consent.

Exclusion Criteria:

* Presence of co-morbidities including cancer, congestive heart failure, connective tissue disease and hematologic diseases;
* Inadequately dialyzed, indicating by urea clearance index (KT/V) < 1.20;
* Presence of severe physical symptoms such as bone pain, itchy skin, sleep apnea and restless legs which are obviously causative for insomnia; and weary condition caused by severe anemia (hemoglobin<60g/L) or malnutrition (serum albumin<30g/L).
* Infections of external ears or malformed ears.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
clinical response rate | at 8 weeks from baseline
  Response is defined as a reduction of Pittsburgh sleep quality index (PSQI) global score by 3 points and more according to literature review

SECONDARY OUTCOMES:
change of PSQI scores at the end of treatment | change from baseline PSQI scores at 8 weeks
  PSQI scores will include PSQI global score, and scores of each domain (i.e. sleep duration, sleep disturbance, sleep latency, day dysfunction, sleep efficiency, overall sleep quality and sleep medication).
change of PSQI scores at the first followup | change from baseline PSQI scores at 12 weeks
  PSQI scores will include PSQI global score, and scores of each domain (i.e. sleep duration, sleep disturbance, sleep latency, day dysfunction, sleep efficiency, overall sleep quality and sleep medication).
change of PSQI scores at the second followup | change from baseline PSQI scores at 16 weeks
  PSQI scores will include PSQI global score, and scores of each domain (i.e. sleep duration, sleep disturbance, sleep latency, day dysfunction, sleep efficiency, overall sleep quality and sleep medication).
change of PSQI scores at the third followup | change from baseline PSQI scores at 20 weeks
  PSQI scores will include PSQI global score, and scores of each domain (i.e. sleep duration, sleep disturbance, sleep latency, day dysfunction, sleep efficiency, overall sleep quality and sleep medication).
weekly dose of hypnotics | Day 0 (baseline), at 8 weeks (the end of treatment), at 12 weeks (the first followup),at 16 weeks (the second followup) and at 20 weeks (the third followup)
  If participants required hypnotic agents during the study because of unbearable sleep disorders, they will be allowed to take hypnotics initiating from the minimum dose and encouraged to complete the trial. The weekly dose of hypnotic agents will be recorded.
adverse events | through study completion, an average of 20 weeks
  Adverse events throughout the treatment and follow-up periods, regardless of its relevance to the interventions, will be documented and dealt with by appropriate measures.

CONTACTS AND LOCATIONS:
Overall Officials: Qizhan Lin, MD, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (6):
- China (6):
  - Guangzhou HEMC (Higher Education Mega Center) Hospital, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Guangzhou Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangzhou Charity Hospital, Guangzhou, Guangdong
  - Wuyi Hospital of Traditional Chinese Medicine, Jiangsu Sheng, Guangdong
  - Shenzhen Hospital of Traditional Chinese Medicine, Shebu, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
IPD including the demographic information, PSQI scores and drug use at baseline and 8,12,16,20 week from baseline of all participants will be shared. The data will be availbale at ResMan® Clinical Trial Management Public Platform, with the link http://www.medresman.org/uc/index.aspx

REFERENCES:
- [Result] Zou C, Yang L, Wu Y, Su G, Chen S, Guo X, Wu X, Liu X, Lin Q. Auricular acupressure on specific points for hemodialysis patients with insomnia: a pilot randomized controlled trial. PLoS One. 2015 Apr 15;10(4):e0122724. doi: 10.1371/journal.pone.0122724. eCollection 2015. PMID 25874938
- [Result] Wu Y, Zou C, Liu X, Wu X, Lin Q. Auricular acupressure helps improve sleep quality for severe insomnia in maintenance hemodialysis patients: a pilot study. J Altern Complement Med. 2014 May;20(5):356-63. doi: 10.1089/acm.2013.0319. Epub 2014 Feb 26. PMID 24571603
- [Derived] Wu Y, Yang L, Zhong Z, Wu X, He Z, Ma H, Cai C, Li Y, Wu X, Fu B, Chen X, Wang L, Zhao D, Meng X, Qi A, Yang A, Li L, Liu X, Zou C, Lin Q. Auricular Acupressure for Hemodialysis Patients with Insomnia: A Multicenter Double-Blind Randomized Sham-Controlled Trial. J Integr Complement Med. 2022 Apr;28(4):339-348. doi: 10.1089/jicm.2021.0332. Epub 2022 Jan 13. PMID 35426736
- [Derived] Wu Y, Yang L, Li L, Wu X, Zhong Z, He Z, Ma H, Wang L, Lu Z, Cai C, Zhao D, Meng X, Qi A, Yang A, Su G, Guo X, Liu X, Zou C, Lin Q. Auricular acupressure for insomnia in hemodialysis patients: study protocol for a randomized controlled trial. Trials. 2018 Mar 7;19(1):171. doi: 10.1186/s13063-018-2546-2. PMID 29514705
- See also: previously finished pilot RCT — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0122724
- See also: observational study on auricular acupressure — http://online.liebertpub.com/doi/abs/10.1089/acm.2013.0319